CLINICAL TRIAL: NCT02562001
Title: Association of Transcranial Direct Current Stimulation (tDCS) With Gait Training With Partial Body Weight Support on the Robotic Device (Lokomat) for Treatment of Patients With Incomplete Spinal Cord Injury
Brief Title: Association Between tDCS and Lokomat Training in Patients With Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Linamara Rizzo Battistella, MD PhD, Professor of the Medical School, USP; Chairman of the Board of Medical and Physical Rehabilitation Institute (IMREA), University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43450715.7.0000.0068_CAAE
Record Dates: First submitted 2015-07-30; First posted 2015-09-29 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; gait training; robotic; Lokomat; Transcranial Magnetic Stimulation; transcranial direct-current stimulation; Electroencephalography; Functional near-infrared spectroscopy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Outpatient active group (Experimental): This group will receive active tDCS, combined with Lokomat gait training
  Interventions: Device: Outpatient active group
- Inpatient active group (Experimental): This group will receive active tDCS, combined with Lokomat gait training
  Interventions: Device: Inpatient active group
- Outpatient placebo group (Experimental): This group will receive placebo tDCS, combined with Lokomat gait training
  Interventions: Device: Outpatient placebo group
- Inpatient placebo group (Experimental): This group will receive placebo tDCS, combined with Lokomat gait training
  Interventions: Device: Inpatient placebo group

INTERVENTIONS:
Device: Outpatient active group — active tDCS during 20 minutes before Lokomat training for outpatients
  Other Names: tDCS active
  Arms: Outpatient active group
Device: Outpatient placebo group — placebo tDCS during 20 minutes before Lokomat training for outpatients
  Other Names: tDCS placebo
  Arms: Outpatient placebo group
Device: Inpatient active group — active tDCS during 20 minutes before Lokomat training for inpatients
  Other Names: tDCS active
  Arms: Inpatient active group
Device: Inpatient placebo group — placebo tDCS during 20 minutes before Lokomat training for inpatients
  Other Names: tDCS placebo
  Arms: Inpatient placebo group

SUMMARY:
The spinal cord injury is identified as the major cause of permanent disability worldwide, with the loss of ability to walk being the largest and most devastating of them for these patients. Our goal is to analyze the effects of electrical transcranial direct-current stimulation (tDCS) combined with gait training with partial body weight support aided by robotic device (Lokomat, Hocoma) in the gait of patients with incomplete spinal cord injury (SCI). In this stratified randomized double-blind study, the participants will be randomly allocated into one of both groups, outpatients (GA) or inpatients (GI), and will receive active or placebo tDCS followed by gait training with Lokomat (GA: 3 sessions/week x 10 weeks = 30 sessions; GI: 5 sessions/week x 6 weeks = 30 sessions). The functional assessments (through clinical and functional scales, assess gait, muscle strength, spasticity, balance and pain) and neurophysiological (cortical excitability measured by transcranial magnetic stimulation, electroencephalography and functional near-infrared spectroscopy) will be held before and after the training period. The functional assessments will be also held after 15 sessions (intermediate) and after 3 months follow up. The expected result is that patients that received the active tDCS presents an improvement over the ground gait after the Lokomat training period significantly greater than the placebo group, with relations between neurophysiologic, kinematics and functional measurements.

DETAILED DESCRIPTION:
The spinal cord injury is identified as the major cause of permanent disability worldwide, with the loss of ability to walk being the largest and most devastating of them for these patients. Therefore, our goal is to analyze the effects of the treatment with electrical transcranial direct-current stimulation (tDCS) associated with gait training with partial body weight support aided by robotic device (Lokomat, Hocoma) in the gait of patients with incomplete spinal cord injury (SCI) classified as AIS C and D. In this stratified randomized double-blind study, the participants will be randomly allocated into one of both groups, outpatients (GA) or inpatients (GI), and will receive active or placebo tDCS followed by gait training with Lokomat (GA: 3 sessions/week x 10 weeks = 30 sessions; GI: 5 sessions/week x 6 weeks = 30 sessions). The functional assessments (through clinical and functional scales, assess gait, muscle strength, spasticity, balance and pain) and neurophysiological (cortical excitability measured by transcranial magnetic stimulation, electroencephalography and functional near-infrared spectroscopy) will be held before and after the training period. The functional assessments will be also held after 15 sessions (intermediate) and after 3 months follow up. The expected result is that patients that received the active (tDCS) presents an improvement over the ground gait after the Lokomat training period, significantly greater than the placebo group, with positive correlation between neurophysiologic, kinematics and functional measurements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of incomplete spinal cord injury of traumatic origin;
* 1 to 36 months of lesion;
* ASIA C and D;
* Stable clinical status;
* Cognitive function preserved in order to understand and execute the experiment and follow the instructions (Wechsler Adult Intelligence Scale - WASI 2014);
* Written informed consent;
* Tolerance to sit upright for at least 1 hour.

Exclusion Criteria:

* Traumatic brain injury history, stroke, epilepsy and/or any other previous or concomitant neurological conditions to spinal cord injury;
* Presence of progressive neurodegenerative disease;
* Previous orthopedic problems (eg osteoarthritis, joint deformities);
* Member hypertonic (grade > 3 on the modified Ashworth scale);
* Active/passive joint range of motion limitations;
* Irreversible muscle contractures;
* Lack of physical resistance during proposed physical training;
* Disabling fatigue;
* Body weight > 150 Kg;
* Osteoporosis with pathological fracture risk;
* Asymmetry in the lower limbs > 2 cm;
* Skin lesions and / or pressure ulcer in areas where the orthosis of Lokomat will press;
* Any other exclusion criteria established by medical decision.

Exclusion criteria for TMS:

Skin lesions in the stimulation site; presence of electric, magnetic or mechanically activated implant (including cardiac pacemakers); intracerebral vascular clip or any other electrically sensitive device; pregnancy; metal in any part of the head; history of epilepsy resistant to medication; history of seizures or loss of consciousness not clarified and / or unaccompanied by a doctor.

Exclusion criteria for Lokomat:

Cardiac pacemaker; unstable angina or other decompensated heart disease; decompensated chronic obstructive pulmonary disease; unchecked autonomic dysreflexia that hinders Lokomat training; unhealed fracture of the bones of the lower limbs; tracheostomy; deformities and stiffness of the hip joint, knee ( ≥ 20° flexion) and ankle ( ≥ 10° plantar flexion).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
A. Change in the Walk Index for Spinal Cord Injury, WISCI II | pre (before treatment) [t0], inter (after 15 sessions) [after 5 weeks GA and after 3 weeks GI], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]

SECONDARY OUTCOMES:
American Spinal Injury Association Impairment Scale - ASIA | pre (before treatment) [t0]
Change in the (Wechsler Adult Intelligence Scale - WASI 2014) | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Ashworth Modified Scale | pre (before treatment) [t0],inter (after 15 sessions) [after 5 weeks GA and after 3 weeks GI], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Berg Balance Test | pre (before treatment) [t0],inter (after 15 sessions) [after 5 weeks GA and after 3 weeks GI], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the 10 meters Walking Test and 6 Minutes Walking test | pre (before treatment) [t0], inter (after 15 sessions) [after 5 weeks GA and after 3 weeks GI], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Time Up and Go Test - TUG | pre (before treatment) [t0], inter (after 15 sessions) [after 5 weeks GA and after 3 weeks GI], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Short Form - 36 Quality of Life Test - SF 36 | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Spinal Cord Independence Measure - SCIM | pre (before treatment) [t0], inter (after 15 sessions) [after 5 weeks GA and after 3 weeks GI], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Lower Extremity Isokinetic Dynamometry | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI]
Change in the Visual Analogic Scale - VAS | pre (before treatment) [t0], inter (after 15 sessions) [after 5 weeks GA and after 3 weeks GI], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Brazilian version of the McGill Pain Questionnaire | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Pressure Algometer | pre (before treatment) [t0], inter (after 15 sessions) [after 5 weeks GA and after 3 weeks GI], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Conditioned Pain Modulation - CPM | pre (before treatment) [t0], inter (after 15 sessions) [after 5 weeks GA and after 3 weeks GI], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Pain-Related Self-Statements Scale - Catastrophizing Subscale (PRSS-Catastrophizing) | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Hospital Anxiety and Depression Scale - HAD | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Beck Depression Inventory | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Patient Health Questionnaire 9 - PHQ 9 | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI] and 3 months follow up [after 22 weeks GA and after 18 weeks GI]
Change in the Transcranial Magnetic Stimulation | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI]
Change in the Functional Near-Infrared Spectroscopy - fNIRS 16 optodes (48 channels) | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI]
Change in the Electroencephalography | pre (before treatment) [t0], post (after treatment) [after 10 weeks GA and after 6 weeks GI]

CONTACTS AND LOCATIONS:
Overall Officials: Linamara Battistella, Md PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto de Medicina Física e Reabilitação, Hospital das Clínicas, Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Pai MYB, Terranova TT, Simis M, Fregni F, Battistella LR. The Combined Use of Transcranial Direct Current Stimulation and Robotic Therapy for the Upper Limb. J Vis Exp. 2018 Sep 23;(139):58495. doi: 10.3791/58495. PMID 30295660
- [Result] Simis M, Uygur-Kucukseymen E, Pacheco-Barrios K, Battistella LR, Fregni F. Beta-band oscillations as a biomarker of gait recovery in spinal cord injury patients: A quantitative electroencephalography analysis. Clin Neurophysiol. 2020 Aug;131(8):1806-1814. doi: 10.1016/j.clinph.2020.04.166. Epub 2020 May 22. PMID 32540720